CLINICAL TRIAL: NCT03291015
Title: Kienbock Disease Radiographic Guided Treatment Versus Arthroscopic Guided Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youssef Abdelmalak, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kienbock disease
Record Dates: First submitted 2017-09-07; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Kienbock Disease
Keywords: arthroscopy; radiographic(plain X ray)
MeSH Terms: conditions — Osteonecrosis | interventions — Arthroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiographic guided treatment (Other): radiographic guided treatment of kienbock disease using plain x ray for determine treatment plan
  Interventions: Device: radiographic
- arthroscopic guided treatment (Other): arthroscopic guided treatment of kienbock disease using wrist arthroscopy for determine treatment plan (Wrist arthroscopy)
  Interventions: Device: arthroscopy

INTERVENTIONS:
Device: radiographic — using plain x ray to determind the treatment plan
  Arms: radiographic guided treatment
Device: arthroscopy — using wrist arthroscopy to determind the treatment plan
  Arms: arthroscopic guided treatment

SUMMARY:
To Compare Between Radiological Guided Treatment And Arthroscopic Guided Treatment Of KIENBOCK Disease

DETAILED DESCRIPTION:
Kienbock'sdisease is defined as avascular necrosis of the lunate bone, which may ultimately progress to lunate sclerosis, collapse, and wrist instability. Incidence is highest in males 20-40 years of age, although it may occur in any age group. Kienbock's disease is uncommon in skeletally immature patients. The cause of Kienbock's disease is likely multi factorial, but potential risk factors have been identified including variant lunate arterial supply and ulnar negative variance. In fewer than 20% of patients, the dorsal blood supply is absent and the lunate is supplied by the palmar radiocarpal arch only; this may represent a risk factor for Kienbock's disease .

Negative ulnar variance may also predispose to Kienbock's disease due to abnormal force loading on the lunate.

Kienbock's disease may be staged according to radiologic appearance using Lichtman classification Stage I is defined as normal radiographic appearance of the lunate with marrow edema present on MRI.

In Stage II disease, there is sclerosis of the lunate, with or without a fracture line, but without lunate collapse.

Stage III, defined as presence of lunate articular surface collapse, may be divided further into three subcategories.

In Stage IIIA, there is no scaphoid rotation; in Stage IIIB, there is fixed scaphoid rotatory subluxation, and in Stage IIIC, a coronal fracture of the lunate is present in addition to scaphoid rotation. Stage III C in 2010 as an addition to the classification scheme.

Stage IV disease is present when secondary radiocarpal or midcarpal osteoarthritis is present in addition to Stage III findings.

An alternate classification of Kienbock's disease, the Bain and Begg

The assessment and management of Kienböck Disease (KD) has always been conundrum. The Lichtman classification has traditionally been used to guide treatment based on imaging. Arthroscopy provides a direct visualization of the articular surface,allows probing of the surfaces, and enables minimally invasive techniques to be performed. The Lichtman-Bain classification is a new classification that takes into account the osseous, vascular, and cartilage aspects of the lunate and the secondary effects on the wrist. It identifies the important prognostic factors including age, the status of the lunate, and the status of the wrist.

With arthroscopy, the articular surfaces of the lunate can be assessed to better understand the status of the lunate. The lunate can be defined as intact, compromised,or not reconstructable. If the lunate is intact then lunate decompression (forage) and arthroscopic assisted bone grafting can be performed. If the lunate facet and capitate are functional, then proximal carpectomy can be performed.

Assessment of the wrist includes assessment of the adjacent articular surfaces of the central column articulations (radiocarpal and midcarpal articulations). Instability of the proximal carpal row can also be assessed. The radioscaphoid articulation is often preserved except in late KD, which allows the scaphocapitate fusion to be a good surgical option. This can now be performed as an arthroscopic procedure. Once the radioscaphoid articulation is degenerate, a salvage procedure is required Wrist arthroscopy is a commonly used procedure that has undergone many modifications and improvements since it was first described. The advent of new portals (both dorsal and volar) means that the wrist joint can be viewed from virtually any perspective ("box concept"). Indications for wrist arthroscopy have continued to expand and include diagnostic and reparative procedures and, more recently, reconstructive, soft-tissue, and bony procedures. Arthroscopic grading of Kienböck's disease better describes articular damage compared with plain radiographs and can help guide surgical treatment options This grading system assists in classifying the severity of the disease and better directs the surgeon toward the reconstructive surgical options grade 0 disorder could be treated with an extra-articular procedure, such as a joint-leveling procedure or revascularization of the lunate. Patients with grade 1or 2a can be treated with a radio-scapho-lunate fusion Patients with grade 1 or 2b can be treated with aproximal-row carpectomy, whereas those with grade 3or 4 require salvage procedures (such as wrist arthrodesis or arthoplasty) Menth-Chiari et al.15 reported on the use of arthroscopic debridement for Kienböck's disease. They reportedexcellent pain relief and improved range of motion in all grades of patients with up to 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons with average age of 20-60 years.
* Persons coming to outpatient clinic and trauma unit complaining Of Chronic Wrist pain
* Plain x-ray films Antero-posterior View And lateral views of the Wrist

Exclusion Criteria:

* Persons < 20 years or > 60 years.
* Traumatic WristWithFracture
* Previous Wrist surgery.
* Patient With Condraindication To plain X-Ray

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison Between Radiological Guided Treatment(15Patient) And Arthroscopic Guided Treatment(Other 15Patient) Of KIENBOCK Disease | baseline
  it is found tht 70% ofkienbock disease patient treated by radiographic guided treatment plan is not satisfied sothat we will analyse the persentage of satisfied patient treated by arthroscopic guided treatment plan versus radiographic guided treatment plan

REFERENCES:
- [Background] Nealey EM, Petscavage-Thomas JM, Chew FS, Allan CH, Ha AS. Radiologic Guide to Surgical Treatment of Kienbock's Disease. Curr Probl Diagn Radiol. 2018 Mar-Apr;47(2):103-109. doi: 10.1067/j.cpradiol.2017.04.012. Epub 2017 Apr 25. PMID 28619441
- [Background] Lichtman DM, Lesley NE, Simmons SP. The classification and treatment of Kienbock's disease: the state of the art and a look at the future. J Hand Surg Eur Vol. 2010 Sep;35(7):549-54. doi: 10.1177/1753193410374690. Epub 2010 Jul 9. PMID 20621943
- [Background] Stahl S, Stahl AS, Meisner C, Hentschel PJH, Valina S, Luz O, Schaller HE, Lotter O. Critical analysis of causality between negative ulnar variance and Kienbock disease. Plast Reconstr Surg. 2013 Oct;132(4):899-909. doi: 10.1097/PRS.0b013e31829f4a2c. PMID 24076682
- [Background] Roth JH, Poehling GG, Whipple TL. Arthroscopic surgery of the wrist. Instr Course Lect. 1988;37:183-94. PMID 3418121
- [Background] Bain GI, Munt J, Turner PC. New advances in wrist arthroscopy. Arthroscopy. 2008 Mar;24(3):355-67. doi: 10.1016/j.arthro.2007.11.002. Epub 2008 Jan 29. PMID 18308189
- [Background] Bain GI, Begg M. Arthroscopic assessment and classification of Kienbock's disease. Tech Hand Up Extrem Surg. 2006 Mar;10(1):8-13. doi: 10.1097/00130911-200603000-00003. PMID 16628114
- [Background] Bain GI, MacLean SB, Tse WL, Ho PC, Lichtman DM. Kienbock Disease and Arthroscopy: Assessment, Classification, and Treatment. J Wrist Surg. 2016 Nov;5(4):255-260. doi: 10.1055/s-0036-1584546. Epub 2016 Jun 20. PMID 27777814
- [Background] Bain GI, Durrant A. An articular-based approach to Kienbock avascular necrosis of the lunate. Tech Hand Up Extrem Surg. 2011 Mar;15(1):41-7. doi: 10.1097/BTH.0b013e31820e82e8. PMID 21358525